CLINICAL TRIAL: NCT03623204
Title: Evolution of Dyspnea After Bariatric Surgery in Patient With Obesity
Acronym: OBES-DYSP
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2017Ao007
Record Dates: First submitted 2018-08-07; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Obesity
Keywords: Obesity; Dyspnea; Bariatric Surgery
MeSH Terms: conditions — Obesity; Dyspnea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with bariatric surgery for obesity
  Interventions: Other: Dyspnea evaluation

INTERVENTIONS:
Other: Dyspnea evaluation

SUMMARY:
Obesity, defined as a Body Mass Index greater than or equal to 30 kg/m2, represents a significant public health issue. Dyspnea is a very common and crippling symptom in obesity. About 80% of people with obesity experience dyspnea in daily living. Bariatric surgery has been demonstrated to be an excellent treatment for obesity by inducing significant weight loss. Nevertheless, changes in dyspnea in daily living after bariatric surgery and the links between variations in dyspnea and lung function tests after bariatric surgery have not been previously investigated.

DETAILED DESCRIPTION:
The objective of this study was to determine if bariatric surgery is associated with an improvement of dyspnea in daily living according to the mMRC scale in patients with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Obesity
* scheduled bariatric surgery

Exclusion Criteria:

- age < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with obesity and who underwent bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2016-02-01 (Actual)

PRIMARY OUTCOMES:
Dyspnea in daily living evaluated using the mMRC scale | Month 6
  Dyspnea in daily living evaluated using the mMRC scale
Dyspnea in daily living evaluated using the mMRC scale | Month 12
  Dyspnea in daily living evaluated using the mMRC scale

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France

REFERENCES:
- [Background] Boissiere L, Perotin-Collard JM, Bertin E, Gaubil I, Diaz Cives A, Barbe C, Dury S, Nardi J, Lebargy F, Deslee G, Launois C. Improvement of dyspnea after bariatric surgery is associated with increased Expiratory Reserve Volume: A prospective follow-up study of 45 patients. PLoS One. 2017 Sep 20;12(9):e0185058. doi: 10.1371/journal.pone.0185058. eCollection 2017. PMID 28931052